CLINICAL TRIAL: NCT05997004
Title: Glycopyrrolate Prophylaxis for Prevention of Bradyarrhythmia During Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Academy of Medical Sciences, Nepal (Other Government)
Responsible Party: Principal Investigator, Brihaspati K C, Principal Investigator, National Academy of Medical Sciences, Nepal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NAMS Nepal
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Bradyarrhythmia; Cardiac Arrest; Tachycardia; Asystole
Keywords: Glycopyrrolate; Bradyarrhythmia; Laparoscopy; Pneumoperitoneum; Cardiac Arrest
MeSH Terms: conditions — Bradycardia; Heart Arrest; Tachycardia; Pneumoperitoneum | interventions — Saline Solution; Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to two groups having 31 in each, by using a computer-generated table of random numbers which was enclosed in a sealed envelope and was opened by an anesthesiologist who were not involved in the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): 31 participants received 1ml of Normal Saline
  Interventions: Drug: Normal Saline
- Glyco (Experimental): 31 participants received 1ml (0.2mg) of Glycopyrrolate
  Interventions: Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Normal Saline — After surgical creation of umbilical port Control group received injection normal saline 1ml.
  Arms: Control
Drug: Glycopyrrolate — After surgical creation of umbilical port Group II received injection Glycopyrrolate 1ml=0.2mg
  Arms: Glyco

SUMMARY:
The goal of this clinical trial is to evaluate the incidence of bradycardia during laparoscopic cholecystectomy. The main question[s] it aims to answer are:

* Does bradycardia really occurs during pneumoperitoneum/laparoscopic surgery?
* If the patient get Glycopyrrolate, Does it really prevent pneumoperitoneum/laparoscopic surgery induced bradycardia?

DETAILED DESCRIPTION:
The emergence of laparoscopic surgery has changed the way of approach for several organs. Despite several advantages, laparoscopic surgery may result in serious complications due to the physiologic changes which occur during the procedure. The cardiovascular system is one of the most challenged systems of the human body during laparoscopy. The insufflation of gas into the peritoneal cavity can provoke arrhythmias. Their incidence is as high as 14-27% of laparoscopies which is higher than in 'open' surgery. The life-threatening bradyarrhythmia (sinus bradycardia, nodal rhythm, atrio-ventricular dissociation and asystole) are frequently encountered during laparoscopic procedure which are due to a vagal-mediated cardiovascular reflex initiated by rapid stretching of the peritoneum at the beginning of peritoneal insufflation. There are studies addressing measures to prevent or control cardiovascular catastrophes during laparoscopic cholecystectomy. Some studies suggest administration of anticholinergic agents especially glycopyrrolate and atropine for prevention of bradycardia during intra-abdominal laparoscopic surgeries. Whereas some study suggests judicious use of Atropine as it increases the risk of tachyarrhythmia. Glycopyrrolate is a synthetic anticholinergic commonly used as a preoperative antimuscarinic agent to reduce salivary, tracheobronchial, and pharyngeal secretions, to reduce the volume and free acidity of gastric secretions, and to block cardiac vagal inhibitory reflexes during induction of anesthesia and intubation.

HYPOTHESIS Glycopyrrolate administration reduces the incidence of bradycardia during Laparoscopic Cholecystectomy.

General objectives To evaluate the role of Glycopyrrolate on prevention of bradyarrhythmia during Laparoscopic cholecystectomy.

Specific objective

1. To evaluate the change in heart rate and rhythm at different time interval after pneumoperitoneum.
2. To evaluate the change in Systolic, diastolic and Mean arterial blood pressure at different time interval after pneumoperitoneum.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of either sex aged 15-65 years
2. Patient undergoing elective laparoscopic cholecystectomy
3. American Society of Anesthesiologists (ASA) physical status I

Exclusion Criteria:

1. Patients with history of recent or past cardiac diseases
2. Patients with pre-operative heart rate ≤60beats/min.
3. Patients on cardiac medications
4. Allergic to Glycopyrrolate

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Heart Rate (Bradycardia) | Starting at 1minutes after creation of pneumoperitoneum up to Extubation (Recorded at 1,3,5,10,20,30,40,50 minutes after pneumoperitoneum and before and after extubation)
  The primary outcome will be Bradycardia defined as heart rate below 60beats per minute

SECONDARY OUTCOMES:
Systolic Blood Pressure | Starting at 1minutes after creation of pneumoperitoneum up to Extubation (Recorded at 1,3,5,10,20,30,40,50 minutes after pneumoperitoneum and before and after extubation)
  Monitoring of systolic Blood pressure
Diastolic Blood Pressure | Starting at 1minutes after creation of pneumoperitoneum up to Extubation (Recorded at 1,3,5,10,20,30,40,50 minutes after pneumoperitoneum and before and after extubation)
  Monitoring of diastolic Blood pressure
Mean Arterial Pressure | Starting at 1minutes after creation of pneumoperitoneum up to Extubation (Recorded at 1,3,5,10,20,30,40,50 minutes after pneumoperitoneum and before and after extubation)
  Monitoring of Mean Arteria pressure

CONTACTS AND LOCATIONS:
Overall Officials: Brihaspati K C, MD, Principal Investigator — NAMS Bir Hospital; Brahmadev Jha, MD, Study Chair — NAMS Bir Hospital; Surendra Bhusal, MD, Study Chair — NAMS Bir Hospital
Locations (1):
- National Academy of Medical Sciences, Kathmandu, Nepal